CLINICAL TRIAL: NCT06825949
Title: A Phase II Single-Arm Clinical Study to Explore the Efficacy and Safety of Hyperbaric Oxygen in the Neoadjuvant Treatment of Hormone Receptor Positive Breast Cancer Patients
Brief Title: A Clinical Study to Explore the Efficacy and Safety of Hyperbaric Oxygen in the Neoadjuvant Treatment of Hormone Receptor Positive Breast Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Kun Wang, Professor, Guangdong Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2024-1084-02
Record Dates: First submitted 2025-01-21; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancers
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hyperbaric Oxygen group (Experimental): Patients who meet the inclusion criteria will be enrolled and given hyperbaric oxygen intervention, with a minimum of 5 times hyperbaric oxygen treatments per chemotherapy cycle, one per day for 60-90 minutes, for a total of 30-40 hyperbaric oxygen treatments (100% oxygen at a pressure of 2.0 ATA).
  Interventions: Device: Hyperbaric oxygen treatment

INTERVENTIONS:
Device: Hyperbaric oxygen treatment — Patients who meet the inclusion criteria will be enrolled and given hyperbaric oxygen intervention, with a minimum of 5 hyperbaric oxygen treatments per chemotherapy cycle, one per day for 60-90 minutes, for a total of 30-40 hyperbaric oxygen treatments (100% oxygen at a pressure of 2.0 ATA).

SUMMARY:
The goal of this study is to explore the efficacy and safety of hyperbaric oxygen in the neoadjuvant treatment of hormone receptor positive breast cancer patients

ELIGIBILITY:
Inclusion Criteria:

1. understood the study process, volunteered to participate in this study and signed an informed consent form
2. Patients with histopathologically confirmed diagnosis of initial unilateral primary invasive breast cancer, occult breast cancer, Inflammatory breast cancer and eczema-like carcinoma are excluded.
3. Female, aged ≥ 18 years and ≤ 60 years.
4. Patients who meet the inclusion criteria of neoadjuvant therapy to receive neoadjuvant therapy for breast cancer (locally advanced breast cancer (AJCC Stage III, except T3N1M0), or operable, but do not meet the conditions of breast conservation or axillary preservation (Stage IIA-IIB and T3N1M0).
5. Hormone receptor-positive breast cancer (Luminal/HER2-low (IHC 2+/FISH-negative)).
6. ECOG performance status 0-1.
7. LVEF ≥ 55 per cent
8. Adequate bone marrow functional reserve: white blood cell count ≥ 3.0 x 109/L, neutrophil count ≥ 1.5 x 109/L; platelet count ≥ 100 x 109/L; haemoglobin ≥ 90g/L;
9. AST, ALT ≤ 2.5 times the upper limit of normal value, alkaline phosphatase ≤ 2.5 times the upper limit of normal value, total bilirubin ≤ 1.5 times the upper limit of normal value; serum creatinine ≤ 1.5 times the upper limit of normal value
10. For non-menopausal or non-surgically sterilised female patients: consent to contraception during treatment and for at least 7 months after the last dose of study treatment

Exclusion Criteria:

1. have contraindications to hyperbaric oxygen therapy: lung disease (severe chronic obstructive airway disease, herpetic lung disease, acute or chronic lung infections, uncontrolled asthma, untreated pneumothorax), previous history of middle ear surgery, middle ear disease (eustachian tube dysfunction\recurrent vertigo), eye disease (retinal detachment).
2. Previous hyperbaric oxygen therapy.
3. Distant metastases, including lymph node metastases in the contralateral breast and mediastinum.
4. Malignancy other than radically treated basal or squamous cell carcinoma of the skin or CIS of the uterine cervix within the last two years.
5. Pregnancy or lactation.
6. Uncontrolled hypertension, cardiac, hepatic, renal related diseases or other medical or psychiatric disorders.
7. Major surgical procedures unrelated to breast cancer within 4 weeks prior to randomisation, or patients who have not fully recovered from such surgical procedures.
8. Serious or uncontrolled infections that may interfere with study treatment or assessment of study results, including but not limited to active hepatitis virus infection, human immunodeficiency virus (HIV) antibody positivity, pulmonary infection, or other infections.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
RCB 0/1 rate | After completion of standard cycle of neoadjuvant therapy (through study completion, an average of half a year)

SECONDARY OUTCOMES:
pCR rate after hyperbaric oxygen combined with neoadjuvant therapy in breast cancer patients | After completion of standard cycle of neoadjuvant therapy (through study completion, an average of half a year)
The Miller and payne classification | After completion of standard cycle of neoadjuvant therapy (through study completion, an average of half a year)
RECIST criteria | After completion of the first cycle of adjuvant therapy, After completion of standard cycle of neoadjuvant therapy (through study completion, an average of half a year)
Life quality (EORTC QLQ C-30、EORTC QLQ BR-23 questionnaire) | At the time of patient enrolment, Each cycle of chemotherapy (8 cycle, each cycle is 3 weeks) , Day before surgery, 3 months after surgery
Side effects of hyperbaric oxygen therapy | during the hyperbaric oxygen therapy (up to half a year)
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | through study completion ( an average of half a year)
the Tumor immune microenvironment of the Hyperbaric Oxygen Therapy and neoadjuvant therapy | the time when the patient enrollment, at the end of the first cycle of neoadjuvant therapy (at about the first month) , surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China